CLINICAL TRIAL: NCT01912261
Title: Phase III Randomized Double Blind Placebo-Controlled Study To Assess The Effects Of FeraMax When Administered Orally Once A Day On Postoperative Fatigue Levels In Patients Following Elective Coronary Artery Bypass Graft Surgery (CABG)
Brief Title: Effects of Oral Iron on Postoperative Fatigue Upon Coronary Artery Bypass Graft Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was stopped due to time constraints and resources
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Capital Health, Canada (Other); Dalhousie University (Other)
Responsible Party: Principal Investigator, Blaine Kent MD, Anethesiology, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TheEffectsofOral Iron052013
Record Dates: First submitted 2013-07-29; First posted 2013-07-31 (Estimated); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Fatigue
Keywords: Coronary artery bypass grafting; Anemia; Postoperative fatigue; Functional Capacity; Iron; Adherence; Quality of Life
MeSH Terms: conditions — Fatigue; Anemia | interventions — Sugars; Niferex

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FeraMax (Active Comparator): FeraMax Polysaccharide iron complex oral iron supplement 150mg one capsule orally daily
  Interventions: Drug: Polysaccharide iron complex
- Placebo (Placebo Comparator): one capsule orally daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — one capsule orally daily times 84 days
  Other Names: Sugar pill
  Arms: Placebo
Drug: Polysaccharide iron complex — 150 mg daily orally times 84 days
  Other Names: FeraMAX
  Arms: FeraMax

SUMMARY:
The purpose of this research study is to examine how an oral iron supplement (Feramax®) influences fatigue during early postoperative recovery (at three months) among CABG patients and, the effects on recovery outcomes (e.g. quality of life, functional capacity, anemia, and medication adherence).

It is hypothesized that CABG surgery patients receiving oral iron (Feramax®) 150mg orally (once a day therapy) will have a 15% reduction in POF (measured by the Identity Consequence Fatigue Scale (ICFS)), compared to patients receiving a placebo.

DETAILED DESCRIPTION:
Postoperative fatigue (POF) is one of the main complaints in approximately 39-80% of CABG surgery patients. POF can have a significant impact on an individual's quality of life (QoL) and recovery. The objectives are to examine how an oral iron (Feramax®) influences fatigue during early postoperative recovery (at three months) among CABG patients and determine the effects on recovery outcomes (e.g. QoL, functional capacity, anemia, and medication adherence). To achieve these objectives the research will aim to answer the following questions:

1. Is oral iron effective in reducing POF measured by the Identity Consequence Fatigue Scale (ICFS) over 12 weeks?
2. If oral iron is effective, how effective was it on improving fatigue, functional capacity, QoL, and anemia?
3. To what degree do patients taking oral iron adhere to the prescription? A prospective, randomized, double-blind placebo-controlled, single-center study was chosen for this study. Three hundred participants who are scheduled for an isolated CABG surgery will be recruited from the QEII Health Sciences Centre (QEIIHSC), Halifax, Nova Scotia. All study participants will be followed for three months following hospital discharge.

Data will be collected at five time points:

Time point 1 Baseline -Patients are screened in the preadmission clinic or nursing unit and recruited for the study. During this visit, the patient will be assessed for eligibility, demographic data and blood work collected and three questionnaires and six minute walk test completed by participants.

Time point 2 Discharge/Randomization-Patients will be randomized to either FeraMAX® or placebo at hospital discharge. The treatment will be taken once daily for 84 days starting Day 1 (day after discharge from hospital). The questionnaires, six minute walk test and blood work will be repeated.

Time point 3 -Post testing 7 to 14 days post discharge A follow up telephone call to reminder patients to take medications and fill put side effects diary

Time Point 4 Six week Follow up-Blood work will be collected and three questionnaires and six minute walk test completed by participants.

Time Point 5-End of treatment-The questionnaires, six minute walk test, blood work, collect side effects diary and pill count will be repeated during a clinic visit.

Fatigue will be measured with the ICFS and Functional Assessment of Cancer Therapy Anemia( FACT-An) questionnaire. The Short Form-36 is used to measure QoL and the six minute walk test to measure functional capacity. Standard of care laboratory tests including (hemoglobin (Hgb) level, reticulocyte count, ferritin, iron, total iron binding capacity (TIBC), transferrin saturation, and C-Reactive Protein levels will be drawn. Medication adherence to the will be assessed by pill count.

The primary endpoint will be analyzed using ANOVA for repeated measures to compare level of fatigue of two groups at baseline, discharge, six weeks and 12 weeks. For the secondary endpoint, a subgroup analysis will be performed and reported on participants with and without iron- deficiency anemia to determine if any efficacy of iron on POF is restricted to this population or to a more general population post CABG surgery. Results will be reported using mean and standard deviation when appropriate and median (interquartile range) for nonparametric data. Categorical variables will be compared using Fisher exact test or t test when appropriate. Level of significance was set at p < 0.05.

Oral iron is inexpensive and effective treatment for iron deficiency that occurs from surgical blood loss. Currently there is no specific drug used to treat POF. Standard of care for POF consists of treating and eliminating the underlying symptoms.

ELIGIBILITY:
Inclusion Criteria:

• Non-Urgent, first time, coronary artery bypass grafting.

* American Society of Anesthesia (ASA) physical status II-IV
* Aged 19 years and older
* Able to make informed consent by understanding the nature of the participation
* Able to read and write English to the degree necessary to participate in interviews and questionnaires

Exclusion Criteria:

* Had prior median sternotomy surgery
* A Hemoglobin greater than or equal 120g/L at discharge
* Previous history of noncompliance with oral medications
* Received erythropoiesis-stimulating agents (e.g. epoetin alfa and darbepoetin alfa) postoperatively to discharge
* Allergy to iron History of hematological disorders that are deemed clinically significant as per the investigator's clinical judgment
* Received Clopidogrel within two days prior to surgery, greater than 81mg of Acetylsalicylic acid 24 hours prior to surgery, or have received "new oral anticoagulants" (e.g. Apixaban, Rivaroxaban, and Dabigatran) within the recommended preoperative exclusion period
* History of iron metabolism disorders e.g. known iron overload, hemochromatosis, porphyria
* Chronic fatigue syndrome (a condition that is distinguished from other types of fatigue by fatigue lasting more than six months and has at least four other symptoms (e.g. sleep disturbances, headaches, joint pain, and concentration difficulties) that could contribute to increased fatigue (Afari & Buchwald, 2003)).
* A serum transferrin saturation of more than 50% at discharge
* History of Fibromyalgia
* Current diagnosis of depressive disorder
* History of Hypothyroidism includes uncontrolled thyroid disease (abnormal Thyroid Stimulating Hormone (TSH) or Thyroxine (T4) at screening visit) as per the Investigator's clinical judgment
* Patient taking iron supplementation ≤ 60 days before surgery and in the postoperative period
* Any other unstable conditions as per the Investigator's clinical judgment
* Contraindications to the six-minute walk test
* Physical disability preventing safe performance
* Resting heart rate > 120 beats/min 10 min after rest (relative contraindications)
* Systolic blood pressure >180mm ± Diastolic blood pressure > 100mm Hg (relative contraindications)
* Resting Sp02 <85% on room air or on a prescribed level of supplemental oxygen

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2014-12-16 (Actual); Primary Completion 2018-02-21 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Fatigue Level | 12 weeks after surgery
  Identity Consequence Fatigue scale

SECONDARY OUTCOMES:
Health Related Quality of Life | 12 weeks after discharge from hospital
  Self Report Scale Medical Outcomes Study short Form 36 to measure Quality of Life
Anemia | 12 week after surgery
  Functional Assessment of Cancer Therapy - Anemia Version 4 and Hemoglobin levels
Functional Capacity | 12 weeks after surgery
  Six Minute Walk Test
Medication Adherence | 12 weeks after surgery
  Pill Count

CONTACTS AND LOCATIONS:
Overall Officials: Blaine Kent, MD, Principal Investigator — Capital Health, Canada
Locations (1):
- Capital Health, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No